CLINICAL TRIAL: NCT03618342
Title: Serum Metabolomics Study of Polycystic Ovary Syndrome Based on Liquid Chromatography-Mass Spectrometry
Brief Title: Serum Metabolomics Study of Polycystic Ovary Syndrome
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Heilongjiang University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yan Li, Doctor, Heilongjiang University of Chinese Medicine
Other Study IDs: Metabolomics PCOS
Record Dates: First submitted 2018-08-01; First posted 2018-08-07 (Actual); Last update posted 2020-03-23 (Actual); Status verified 2020-03

CONDITIONS: Polycystic Ovary Syndrome
MeSH Terms: conditions — Polycystic Ovary Syndrome

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- PCOS: PCOS women
- Healthy controls: Healthy control women

SUMMARY:
Polycystic ovary syndrome (PCOS) is a complex, heterogeneous disorder, which produces in 5-20% reproductive age women. In this study, a nontargeted metabolomics approach based on ultra high-performance liquid chromatography coupled with quadrupole time-of-flight mass spectrometry will be used to investigate serum metabolic characteristics of PCOS. PCOS women and healthy control will be divided into two distinct groups based on multivariate statistical analysis. The findings of this study will offer a new insight to understand the pathogenesis mechanism, and the discriminating metabolites may provide a prospect for PCOS diagnosis.

ELIGIBILITY:
Inclusion Criteria:

* PCOS diagnostic criteria: According to the diagnostic criteria revised by the European Society of Human Reproduction and Embryology and the American Society for Reproductive Medicine at the Rotterdam in 2003,4 PCOS patients can be diagnosed if two of the three criteria are present after excluding congenial adrenal hyperplasia, Cushing's syndrome, androgen secreting tumors, or other related disorders. The three criteria are (1) oligo- and/or anovulation; (2) clinical and/or biochemical signs of hyperandrogenism (clinical manifestations of hyperandrogenism include presence of acne, hirsutism, and androgenic alopecia); (3) polycystic ovaries by ultrasound examination: presence of 12 or more follicles in each ovary measuring 2-9 mm on diameter and/or ovarian volume>10 ml.
* Age between 14 and 40 years
* 2 years after menarche

Exclusion Criteria:

-

Ages: 14 Years to 40 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Study Population: PCOS is a complex disease and its pathogenesis is not clear, but it is believed to be the result from genetic, environmental, and lifestyle interaction. It is relatively clear that PCOS is closely related with hormone abnormality. More and more evidence displayed that insulin signaling pathways are closely related to PCOS. PCOS may also be associated with chronic inflammation and increased level of oxidative stress.
Sampling Method: Probability Sample
Enrollment: 1272 (Actual)
Dates: Start 2018-08-02 (Actual); Primary Completion 2019-08-31 (Actual); Study Completion 2020-03-31 (Estimated)

PRIMARY OUTCOMES:
The fatty acid amides (FAAs) metabolite changes | one year
  The metabolic changes between PCOS and healthy controls

SECONDARY OUTCOMES:
The sulfated steroids metabolite changes | one year
  The metabolic changes between PCOS and healthy controls
The free fatty acid metabolite changes | one year
  The metabolic changes between PCOS and healthy controls

CONTACTS AND LOCATIONS:
Locations (1):
- First Affiliated Hospital, Heilongjiang University of Chinese Medicine, Harbin, Heilongjiang, China